CLINICAL TRIAL: NCT06830538
Title: Prospective Observational Spontaneous Study of Anatomical, Functional and QoL Recovery of Patients Undergoing Corneal Transplantation
Brief Title: Study of the Anatomical and Functional Recovery and Quality of Life of Patients Undergoing Corneal Transplantation
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: OFTAFONTANA_OSS_TC
Record Dates: First submitted 2025-01-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Cornea Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the well-being of patients and clinicl outcomes of the cornea after transplantation

DETAILED DESCRIPTION:
The study aims to evaluate patients affected by corneal diseases who will undergo corneal transplantation.

The evaluation will be carried out pre and post transplantation to evaluate the clinical outcome of the patients and the quality of life and functional anatomical recovery.

ELIGIBILITY:
Inclusion Criteria:

* be eighteen years old
* diagnosis of corneal disease with prescription of surgical treatment of corneal transplantation
* sign the informed consent

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with corneal disease who will undergo corneal transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2035-02-01 (Estimated); Study Completion 2035-02-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical recovery after corneal transplant | postoperatively at 7 days, 30 days, 3 months, and 12 months.
  Anatomical recovery will be assessed by the regularity of the cornea.
Visual-functional recovery after corneal transplant | postoperatively at 7 days, 30 days, 3 months, and 12 months.
  Visus examination

SECONDARY OUTCOMES:
Patients's quality of life | One week before surgery and at seven days, thirty days, three months, six months, one year, two years, three years, and four years after surgery.
  Administration to patients of Health-related SF12 questionnaire
Patients's quality of life | One week before surgery and at seven days, thirty days, three months, six months, one year, two years, three years, and four years after surgery.
  Administration to patients of Schedule for the Evaluation of Individual Quality of Life (SEI-QoL) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Fontana, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy